CLINICAL TRIAL: NCT03430466
Title: Phase II Study to Assess Efficacy, Safety & Immunological Biomarker of Anti PD-L1 Antibody + Anti CTLA-4 Antibody in Combination With Hormone Therapy in Patients With Hormone Receptor Positive HER2-negative Recurrent or Metastatic Breast Cancer
Brief Title: Anti PD-L1 Antibody + Anti CTLA-4 Antibody in Combination With Hormone Therapy in Patients With Hormone Receptor Positive HER2-negative Recurrent or Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruiting was not possible
Sponsor: Kyoto Breast Cancer Research Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: kbcrnb001
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalmab&Tremelimumab&Fulvestrant (Experimental): Durvalmab&Tremelimumab&Fulvestrant
  Interventions: Drug: Durvalmab&Tremelimumab&Fulvestrant

INTERVENTIONS:
Drug: Durvalmab&Tremelimumab&Fulvestrant — Durvalumab and Tremelimumab once in 4 weeks Durvalumab for 13 months Tremelimumab for initial 4 months Fulvestrant : At baseline, then week 2, week 4 and after that every 4 weeks

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of anti PD-L1 antibody + anti CTLA-4 antibody in combination with hormone therapy in patients with hormone receptor positive HER2-negative recurrent or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged >= 20 years at informed consent.
2. Patients who have provided written informed consent themselves.
3. Patients who have metastatic and/or advanced lesion
4. Documentation of ER-positive and/or PR-positive tumor (>=1% positive stained cells).
5. Patients with cancer confirmed to be HER2-negative.
6. Patients with confirmed menopause
7. Patients who have plans of 2nd hormone therapy.
8. Patients with a measurable lesion based on RECIST 1.1
9. Patients with ECOG PS of 0 to 1.
10. Patients without any severe disorder in the major organs.

Exclusion Criteria:

-

Exclusion Criteria:

1. Active or prior documented autoimmune disease within the past 2 years.
2. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab or tremelimumab
3. Patients with central nervous system metastasis
4. Patients with life-threatening disease.
5. Patients with a history of treatment with anti-PD-1, anti-PD-L1, anti-PD-L2 or anti-CTLA-4 antibody drug.
6. Patients who have received live vaccination within 30 days before start of the investigational products.
7. Patients with a past medical history of pneumonia requiring steroid treatment or with a past medical history of interstitial pneumonia.
8. Patients considered ineligible for participation in this study by their attending physicians.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Response rate based on RECIST1.1 | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Kyoto University Hospital, Kyoto, Japan